CLINICAL TRIAL: NCT03733626
Title: Clinical Outcomes Associated With the Use of ViviGen® in Conjunction With Posterolateral Fusion for the Treatment of Lumbar Degenerative Disc Disease
Brief Title: Clinical Outcomes Associated With the Use of ViviGen® for the Treatment of Lumbar Degenerative Disc Disease
Acronym: ViviGen
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Corewell Health East (Other)
Collaborators: DePuy Synthes (Industry)
Responsible Party: Principal Investigator, Jad Khalil MD, Staff physician and Assistant Professor of Orthopaedic Surgery, Corewell Health East
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-158
Record Dates: First submitted 2018-10-30; First posted 2018-11-07 (Actual); Results first posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Lumbar Spondylolisthesis; Degenerative Disc Disease; Degenerative Spondylolisthesis; Lumbar Radiculopathy; Lumbar Spinal Stenosis; Lumbar Disc Disease
MeSH Terms: conditions — Spondylolisthesis; Intervertebral Disc Degeneration; Radiculopathy; Spinal Stenosis; Intervertebral disc disease

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to either: 1) treatment arm where the investigator will use an FDA approved/cleared DePuy Synthes spinal pedicle screw system with ViviGen® Cellular Bone Matrix mixed with cortical/cancellous allograft or the 2) control arm where the investigator use the same DePuy Synthes spinal pedicle screw system with local autologous bone graft mixed with cortical/cancellous allograft. Randomization is 1:1
Who Masked: Participant
Masking Description: Participants will be blinded to the randomization group and which bone graft is used during surgery
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- ViviGen® Cellular Bone Matrix with DePuy Synthes Spinal Pedicle Screw System (Active Comparator): 20 subjects undergoing one or two-level instrumented posterolateral lumbar fusion surgery using ViviGen Cellular Bone Matrix mixed with cortical/cancellous allograft and DePuy Synthes pedicle screw system
  Interventions: Combination Product: ViviGen® Cellular Bone Matrix with DePuy Synthes Spinal Pedicle screw system
- Local Bone Autograft with DePuy Synthes Spinal Pedicle Screw System (Placebo Comparator): 20 subjects undergoing open, one or two-level posterolateral lumbar fusion surgery using local autograft mixed with cortical/cancellous allograft and DePuy Synthes pedicle screw system.
  Interventions: Combination Product: Local Bone Autologous Bone Graft with DePuy Synthes Spinal pedicle screw system

INTERVENTIONS:
Combination Product: ViviGen® Cellular Bone Matrix with DePuy Synthes Spinal Pedicle screw system — ViviGen® is manufactured by LifeNet Health. ViviGen® Cellular Bone Matrix is a formulation of cryopreserved viable cortical cancellous bone matrix and demineralized bone. ViviGen is a Human Cells, Tissues, and Cellular and Tissue-based Product (HCT/P) as defined by the U.S. Food and Drug Administration in 21 CFR 1271.10 and will be used with the FDA approved DePuy Synthes Spinal pedicle screw system for fusion.
  Other Names: ViviGen® Cellular Bone Matrix
  Arms: ViviGen® Cellular Bone Matrix with DePuy Synthes Spinal Pedicle Screw System
Combination Product: Local Bone Autologous Bone Graft with DePuy Synthes Spinal pedicle screw system — Patient's own bone harvested during spinal surgery will be used with the FDA approved DePuy Synthes spinal pedicle screw system to create the fusion.
  Other Names: Local Bone Autologous Bone Graft
  Arms: Local Bone Autograft with DePuy Synthes Spinal Pedicle Screw System

SUMMARY:
The objective of this study is to perform a prospective, randomized, controlled clinical trial to compare radiographic fusion rates and patient reported outcomes, including pain and function preoperatively and postoperatively, using Depuy ViviGen® Cellular Bone Matrix mixed with cortical/cancellous allograft in conjunction with an approved Depuy Synthes pedicle screw system compared to autograft mixed with cortical/cancellous allograft in conjunction with the same DePuy Synthes pedicle screw system used for a one or two - level posterolateral lumbar fusion.

DETAILED DESCRIPTION:
This is a prospective randomized, non-blinded, controlled study. Patients with a diagnosis of degenerative disc disease and/or up to grade I spondylolisthesis and planning to undergo a one or two-level instrumented posterolateral lumbar fusion surgery between L1-S1 will be screened. If eligible and the subject meets all the inclusion criteria and none of the exclusion criteria, the subject will be approached about study participation by the surgeon. If the subject agrees to participate, the consent process will be initiated by the study coordinator. Once the patient has been consented; data including medical history, neurological exam, patient questionnaires (visual analogue pain score (VAS), Oswestry low-back disability questionnaire (ODI), short form health survey (SF-36)) will be collected. Randomization will occur once a surgery date has been scheduled so the appropriate instrumentation can be boarded accordingly. A randomization envelope will reveal randomization treatment group. The envelopes will be generated in a 1:1 fashion and be randomly allocated to an assigned study identification number.

Subjects will be randomized to either: 1) treatment arm where the investigator will use an FDA approved/cleared DePuy Synthes spinal pedicle screw system with ViviGen® Cellular Bone Matrix mixed with cortical/cancellous allograft or the 2) control arm where the investigator use the same DePuy Synthes spinal pedicle screw system with local autologous bone graft mixed with cortical/cancellous allograft. Both treatment groups represent standard of care lumbar fusion surgeries using two types of bone graft options to create the arthrodesis as comparators.

Once the lumbar fusion surgery has taken place as planned; data will be collected regarding the surgery performed, including operative time, amount of bone graft used, spinal system used, length of hospital stay, and adverse events/complications.

Study subjects will be followed up at 6-weeks, 3-months, 6-months, and 12-months postoperatively at the private practice or clinic. During these routine (standard of care) postoperative visits, subjects will complete questionnaires (VAS, ODI, SF-36, patient satisfaction) and have neurological exam (lumbar spine exam, see appendix 1) completed by the investigator. Adverse events related to device and/or procedure will be evaluated as each postoperative visit. Anteroposterior (AP) and lateral x-rays will be performed at all visits with flexion and extension x-rays added at baseline, 3-months, 6-months, and 12-months. A CT scan of the lumbar spine will be performed during the 12-month postoperative time frame at the Beaumont-Royal Oak Imaging Center. Radiographic analysis will be performed and evaluated for fusion status as evidenced by bony bridging, presence of radiolucency, and development of pseudoarthrosis at each follow-up visit.

This study design reflects the current standard of care for lumbar spinal stenosis, degenerative disc disease and lumbar degenerative spondylolisthesis. Lumbar fusion surgery using pedicle screw fixation with autograft and allograft bone grafting options is treatment of choice after conservative (non-surgical) therapies have been implemented and failed.

Addendum:

1. In order to protect the well-being of patients and in compliance with the current state mandated shelter in place order, follow-up visits will be completed via telephone visit by the study coordinator when possible. This includes patient reported outcomes and adverse event reporting. Some parts of the study visit may not be completed over the phone such as lumbar x-rays, neuro exam, and CT scan (at 12-months postop); these missing (or scheduled at a later date) protocol specific items will be noted as a protocol deviation with the reason being due to COVID-19.
2. If a televisit is not possible, the visit may be rescheduled at a later date. Therefore, out of window and missing visits will be recorded as protocol deviations with the reason being due to COVID-19.
3. Subject follow-up visits will be rescheduled in the office once the acute phase of the pandemic has subsided if the study visit is not substantially out of window.
4. Subject enrollment is on hold until the acute phase of the pandemic has subsided but screening will continue.

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years of age
2. Able to provide consent
3. Is undergoing standard of care one or two-level instrumented posterolateral fusion at the level between L1-S1
4. Has diagnosis of spinal stenosis, degenerative disc disease and/or up to Grade 1 spondylolisthesis
5. Requires decompression at intended fusion level (multi-level decompression allowed L1-S1)
6. Has failed 6-weeks or more of conservative, non-operative treatment
7. Has back and/or radicular lumbar symptoms with ODI score of ≥ 30 preoperatively.

Exclusion Criteria:

1. Any prior lumbar fusion surgery
2. Requires fusion of more than two levels
3. Requires an interbody fusion based on relevant diagnoses and factors (such as foraminal stenosis, degree of spondylolisthesis, spinal deformity, disc space collapse, and subject's age) as determined by investigator
4. BMI > 40
5. Active systemic infection or infection at operative site
6. History of an osteoporotic fracture and/or vertebral body fracture
7. Is currently being treated with chemotherapy, radiation, immunosuppression or chronic steroid therapy
8. History of osteoporosis, osteopenia, or osteomalacia that would contraindicate spinal surgery
9. Psychological or physical condition in the opinion of the investigator that would interfere with subject self-assessments
10. History of neurological condition in the opinion of the investigator that may affect lumbar function and pain assessments
11. Subjects with a history of cancer must be disease free for at least 3 years
12. Pregnant, or plans on becoming pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2024-06-25 (Actual); Study Completion 2024-06-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jad G Khalil, MD, Principal Investigator — Corewell Health East
Locations (1):
- William Beaumont Hospital, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Boden SD. Overview of the biology of lumbar spine fusion and principles for selecting a bone graft substitute. Spine (Phila Pa 1976). 2002 Aug 15;27(16 Suppl 1):S26-31. doi: 10.1097/00007632-200208151-00007. PMID 12205416
- [Background] Kim DH, Rhim R, Li L, Martha J, Swaim BH, Banco RJ, Jenis LG, Tromanhauser SG. Prospective study of iliac crest bone graft harvest site pain and morbidity. Spine J. 2009 Nov;9(11):886-92. doi: 10.1016/j.spinee.2009.05.006. Epub 2009 Jun 18. PMID 19540168
- [Background] Betz RR. Limitations of autograft and allograft: new synthetic solutions. Orthopedics. 2002 May;25(5 Suppl):s561-70. doi: 10.3928/0147-7447-20020502-04. PMID 12038843
- [Background] Gazdag AR, Lane JM, Glaser D, Forster RA. Alternatives to Autogenous Bone Graft: Efficacy and Indications. J Am Acad Orthop Surg. 1995 Jan;3(1):1-8. doi: 10.5435/00124635-199501000-00001. PMID 10790647
- [Background] DeCoster TA, Gehlert RJ, Mikola EA, Pirela-Cruz MA. Management of posttraumatic segmental bone defects. J Am Acad Orthop Surg. 2004 Jan-Feb;12(1):28-38. doi: 10.5435/00124635-200401000-00005. PMID 14753795
- [Background] DePuy Synthes. https://www.depuysynthes.com/hcp/spine/products/qs/vivigen-cellular-bone-matrix. Copyright DePuy Synthes 2014-2017. DePuy Synthes Biomaterials Division 1302 Wrights Lane East, West Chester, Pennsylvania 19380.
- [Background] Vaccaro AR, Stubbs HA, Block JE. Demineralized bone matrix composite grafting for posterolateral spinal fusion. Orthopedics. 2007 Jul;30(7):567-70. doi: 10.3928/01477447-20070701-06. PMID 17672157
- [Background] Kang J, An H, Hilibrand A, Yoon ST, Kavanagh E, Boden S. Grafton and local bone have comparable outcomes to iliac crest bone in instrumented single-level lumbar fusions. Spine (Phila Pa 1976). 2012 May 20;37(12):1083-91. doi: 10.1097/BRS.0b013e31823ed817. PMID 22076647

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 2 patients were consented but screen failure prior to randomization, leaving 44 patients at start of study
Groups:
- ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System: 20 subjects undergoing one or two-level instrumented posterolateral lumbar fusion surgery using ViviGen Cellular Bone Matrix mixed with cortical/cancellous allograft and DePuy Synthes pedicle screw system
  ViviGen® Cellular Bone Matrix with DePuy Synthes Spinal Pedicle screw system: ViviGen® is manufactured by LifeNet Health. ViviGen® Cellular Bone Matrix is a formulation of cryopreserved viable cortical cancellous bone matrix and demineralized bone.
Period: Overall Study
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Started | 23 | 21
Completed | 19 | 17
Not Completed | 4 | 4
Not completed — Physician Decision | 4 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System | Total
Number analyzed (Participants) | 19 | 17 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.2 (10.5) | 59.8 (11.3) | 60.5 (6.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 9 | 20
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 19 | 17 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 16 | 14 | 30
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 17 | 36

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Successful Lumbar Fusion Measured Radiographically
Description: Count of participants with successful lumbar bone fusion as measured by CT scan and flexion/extension x-rays at 12-months as evidenced by the following three criteria: bony bridging, no presence of radiolucency and no development of pseudoarthrosis at the treated lumbar level
Time Frame: 12 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 19 | 17
Participants | 13 | 11

2. Secondary Outcome: Visual Analog Scale for Pain
Description: Number of participants achieving equal to or greater than a 2-point decrease in patient reported outcomes as measured by Visual Analog Scale for pain (0-10 point scale, 0 = no pain and 10 = severe amount of pain) from baseline to 12-months, representing a decrease in pain.
Time Frame: 12 months postoperative
Population: 4 subjects in autograft arm and 3 subjects in the ViviGen arm did not have 12 month data.
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 16 | 13
Participants | 13 | 12

3. Secondary Outcome: Change in Oswestry Disability Index for Pain and Function
Description: Number of participants achieving equal to or greater than 15-point decrease in patient reported outcomes as measured by Oswestry Disability Index (0-100 point scale, 0 = least amount of disability, 100 = most severe disability) from baseline to 12-months.
Time Frame: 12 months postoperative
Population: 3 participants in the ViviGen group and 4 participants in the Autograft group did not have 12 month data collected
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 16 | 13
Participants | 13 | 11

4. Secondary Outcome: Change in Short Form Health Survey-36 for Quality of Life: Physical Component Summary
Description: Number of participants achieving equal to or greater than 15-point increase in patient reported quality-of-live outcomes as measured by a composite Physical Component Summary score on the SF-36 (0-100 point scale, 0 = low favorable health state and 100 = most favorable health state) from baseline to 12-months. This Physical Component Summary score is calculated by averaging scores from the Pain, Physical Functioning, Physical Role Limitation, and General Health Perception subscales for each patient at 12 months and at baseline, and calculating a difference. A positive number indicates an increase in physical health, and a negative number indicates a decrease in physical health.
Time Frame: 12 months postoperative
Population: 4 participants in the ViviGen group and 4 participants in the Autograft group did not complete12 month SF-36 data
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 15 | 13
Participants | 12 | 9

5. Secondary Outcome: Neurological Deficit Per Lumbar Spine Neurological Exam
Description: Count of participants with new or worsening neurological (lumbar motor and sensory) deficit as evaluated by lumbar spine neurological exam from baseline through 12 months.
Time Frame: 12 months postoperative
Population: 7 participants in the ViviGen Cellular Bone Matrix arm did not complete the 12 month postoperative visit and no data was collected. 5 participants in the local bone autograft arm did not complete the 12 month postoperative visit and no data was collected.
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 12 | 12
Participants | 2 | 2

6. Secondary Outcome: Count of Participants With Revision Surgery by Month 12
Description: Count of participants with revision surgery by month 12
Time Frame: 12 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 19 | 17
Participants | 0 | 0

7. Secondary Outcome: Count of Participants Developing Pseudoarthrosis by Month 12
Description: Count of participants developing pseudoarthrosis by month 12
Time Frame: 12 months postoperative
Measure: Count of Participants; unit: Participants
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
Number analyzed (Participants) | 19 | 17
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/17
Serious Adverse Events (participants affected / at risk) | 1/19 | 0/17
Other Adverse Events (participants affected / at risk) | 9/19 | 11/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System (N=19) | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System (N=17)
Cardiac vessel occlusion (Cardiac disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ViviGen® Cellular Bone Matrix With DePuy Synthes Spinal Pedicle Screw System (N=19) | Local Bone Autograft With DePuy Synthes Spinal Pedicle Screw System (N=17)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4)
Sacroiliac joint pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pseuroarthrosis L4-5 (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dural Tear, intraoperative (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
neurogenic claudication (Nervous system disorders) | 0 (0) | 1 (1)
cervical radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Lower extremity numbness/weakness (Nervous system disorders) | 1 (1) | 2 (3)
Lower extremity pain (Nervous system disorders) | 1 (1) | 1 (1)
Lower extremity radiculopathy (Nervous system disorders) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
COVID-19 infection (Infections and infestations) | 1 (1) | 0 (0)
Surgical site infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-18): https://cdn.clinicaltrials.gov/large-docs/26/NCT03733626/Prot_SAP_000.pdf